CLINICAL TRIAL: NCT06978556
Title: Comparison of Lens Position and Photopic and Mesopic Visual Acuity After Bilateral Implantation of Two Different Diffractive Multifocal Intraocular Lenses.
Brief Title: Photopic and Mesopic Multifocal IOL Performance
Acronym: MIOLRead
Status: Active, not recruiting | Type: Observational
Sponsor: IROC AG (Other)
Collaborators: AMO Ireland (Unknown)
Responsible Party: Principal Investigator, Theo Seiler, Prof. Dr. med. Dr. rer. nat., IROC AG
Other Study IDs: EMEA202102; IE9970584V (Other Grant/Funding Number: AMO IRELAND, Co. Dublin, Ireland)
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cataract; Presbyopia Correction
Keywords: Cataract; multifocal iol; presbyopia; reading speed
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multifocal IOL 1: bilateral pseudophakia with multifocal IOL 1 (Johnson and Johnson Synergy)
  Interventions: Diagnostic Test: No intervention is subject of the study. Only standard pre- and postoperative data will be evaluated.
- Multifocal IOL 2: bilateral pseudophakia with multifocal IOL 2 (Carl Zeiss Meditec AT Lisa Tri)
  Interventions: Diagnostic Test: No intervention is subject of the study. Only standard pre- and postoperative data will be evaluated.

INTERVENTIONS:
Diagnostic Test: No intervention is subject of the study. Only standard pre- and postoperative data will be evaluated. — No intervention is subject of the study. Only standard pre- and postoperative data will be evaluated. Including data from testing refraction, visual acuity, biometry, tomography, and OCT.

SUMMARY:
Modern cataract surgery has become a refractive procedure. Both, multifocal lens implantation and pseudophakic monovision with monofocal IOLs are effective means to address presbyopia correction after cataract surgery. Historically, diffractive multifocal IOLs have provided improved visual acuity at near and intermediate distances and a greater likelihood of spectacle independence than monofocal IOLs.

The light transmittance ratio of the crystalline lens is high and as a monofocal ocular medium that has the ability to modify its shape and geometric properties according to the focal point. Therefore, it is capable of delivering the exact same light energy to the retina, regardless of the distance of the object. Trifocal IOL designs split the light in three focal points. By varying the height of the diffractive step, the amount of light distributed to near, intermediate and distant foci is adjusted according to pupil aperture. The distribution of light to three different foci includes several potential disadvantages, such as loss of visual acuity in mesopic conditions and a loss of contrast sensitivity. Thus, the visual performance of multifocal IOLs depends on several factors, the addition (add) power is a major determinant of the actual range of clear vision, another factor is the light transmittance characteristics of the lens (e.g., the incorporation of a blue light filter).

As different trifocal IOLs become available, it is important to have information on their characteristics regarding visual acuity in order to be able to recommend an IOL that meets the individualized needs of each patient. In order to provide the patient with a high visual acuity in all promised distances, these IOLs need to be aimed at and achieve emmetropia.

Furthermore, multifocal IOLs need good capsular bag centration, they need to remain as unaffected as possible by capsular bag constriction and remain stable in their axial lens position in order to provide a stable refraction after surgery.

The investigators compare the anterior chamber depth stability as marker for positional stability and haptic buckling between two different diffractive IOL designs, one with C-loop haptics and one with plate haptics. Furthermore, the refractive outcome of these IOLs with different designs is examined in photopic and mesopic conditions, as well as visual acuity results for both IOLs.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 45 years of age and older
2. Able to provide written informed consent and follow study instructions in English or German.
3. Desire for spectacle independence
4. Agreement on clinical decision for planned crystalline lens exchange with multifocal IOL implantation (Standardized femtosecond-laser capsulotomy (diameter 5.3mm))
5. Willing and able to return for scheduled follow-up examinations;

Exclusion Criteria:

1. Prior ophthalmic surgery or trauma
2. Zonular-defects, unstable bag
3. Macular pathologies
4. Excessive irregular astigmatism

6. Pregnancy/lactation 7. Predicted Visual acuity of less than 0.8 decimal 8. Participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation;

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing cataract surgery with multifocal IOL implantation at the study site fulfilling inclusion criteria will be asked to participate in the study. All patients are referred by ophthalmologists or are self-referrals at the study site.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
IOL axial position stability | 1, 3, 6, 12 months
  as measured with a biometry and/or anterior segment device.

SECONDARY OUTCOMES:
refraction | 1, 3, 6, 12 months
  standardized ETDRS charts Optometrist blinded
Visual acuity | 1, 3, 6, 12 months
  Standardized with ETDRS charts for far, intermediate, and far distance visual acuity. Defocus curve.
  Optometris is blinded. Measurement in photopic and mesopic conditions
Reading speed | 3 months
  standardized with iRest test. In photopic and mesopic conditions.
  optometrist is blinded.

CONTACTS AND LOCATIONS:
Overall Officials: Theo Seiler, MD, Principal Investigator — IROC AG
Locations (1):
- IROC, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Only upon reasonable request

REFERENCES:
- [Background] Benyoussef AA, Reboux N, Cochener B. Comparison of Bilateral Reading Performance Among Two Presbyopia-Correcting Intraocular Lenses. J Refract Surg. 2022 Jul;38(7):428-434. doi: 10.3928/1081597X-20220516-02. Epub 2022 Jul 1. PMID 35858191
- [Background] Seiler TG, Wegner A, Senfft T, Seiler T. Dissatisfaction After Trifocal IOL Implantation and Its Improvement by Selective Wavefront-Guided LASIK. J Refract Surg. 2019 Jun 1;35(6):346-352. doi: 10.3928/1081597X-20190510-02. PMID 31185099
- [Background] Cillino G, Casuccio A, Pasti M, Bono V, Mencucci R, Cillino S. Working-age cataract patients: visual results, reading performance, and quality of life with three diffractive multifocal intraocular lenses. Ophthalmology. 2014 Jan;121(1):34-44. doi: 10.1016/j.ophtha.2013.06.034. Epub 2013 Aug 14. PMID 23953097
- [Background] Marques EF, Ferreira TB. Comparison of visual outcomes of 2 diffractive trifocal intraocular lenses. J Cataract Refract Surg. 2015 Feb;41(2):354-63. doi: 10.1016/j.jcrs.2014.05.048. PMID 25661129
- [Background] Martinez-de-la-Casa JM, Carballo-Alvarez J, Garcia-Bella J, Vazquez-Molini JM, Morales L, Sanz-Fernandez JC, Polo V, Garcia-Feijoo J. Photopic and Mesopic Performance of 2 Different Trifocal Diffractive Intraocular Lenses. Eur J Ophthalmol. 2017 Jan/Feb;27(1):26-30. doi: 10.5301/ejo.5000814. PMID 27375069
- [Background] Alio JL, Kaymak H, Breyer D, Cochener B, Plaza-Puche AB. Quality of life related variables measured for three multifocal diffractive intraocular lenses: a prospective randomised clinical trial. Clin Exp Ophthalmol. 2018 May;46(4):380-388. doi: 10.1111/ceo.13084. Epub 2017 Nov 29. PMID 29044974
- [Background] Portney V. Light distribution in diffractive multifocal optics and its optimization. J Cataract Refract Surg. 2011 Nov;37(11):2053-9. doi: 10.1016/j.jcrs.2011.04.038. PMID 22018367
- [Background] Hienert J, Hirnschall N, Ruiss M, Ullrich M, Zwickl H, Findl O. Prospective study to compare axial position stability after fellow-eye implantation of 2 distinct intraocular lens designs. J Cataract Refract Surg. 2021 Aug 1;47(8):999-1005. doi: 10.1097/j.jcrs.0000000000000557. PMID 33577276